CLINICAL TRIAL: NCT05363787
Title: The Effect of Therapeutic Touch Applied to Individuals Aged 65-85 With Chronic Disease, Considering the Circadian Cycle, on Sleep Patterns
Brief Title: The Effect of Therapeutic Touch on Sleep Patterns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KaratayUBS
Record Dates: First submitted 2022-04-28; First posted 2022-05-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-04

CONDITIONS: Therapeutic Adherence; Nurse-Patient Relations; Sleep Disorder
MeSH Terms: conditions — Treatment Adherence and Compliance; Sleep Wake Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effect of therapeutic touch on sleep patterns of elderly patients (Experimental): The important effects of the therapeutic approach made by the researcher to the elderly patients hospitalized in the intensive care unit will be evaluated.
  Interventions: Other: therapeutic touch
- Determining the sleep pattern of the Control Group (No Intervention): It will be evaluated whether there is a change in sleep patterns without intervention in the control group.

INTERVENTIONS:
Other: therapeutic touch — Therapeutic Touch (TT) is an evidence-based holistic treatment method in which universal energy is used intentionally and with compassion for a specific purpose, in order to contribute to one's balance and recovery.In a world dominated by technology, one can lose touch with our inner self. We lose our intuitive abilities for beautiful everyday sensations of nature, the surrounding environment, and various visual and auditory elements. The Therapeutic Touch is an ancient Ayurvedic self-massage technique that connects your body to your soul.It is also used in therapeutic communication. Therapeutic communication is the process of influencing and being influenced by one another. It consists of individual-centered, purposeful, planned, effective and satisfying actions.
  Arms: The effect of therapeutic touch on sleep patterns of elderly patients

SUMMARY:
The aim of this study is to determine the effect of the therapeutic touch applied to the sleep patterns of individuals aged 65-85 years with chronic diseases who are treated in the Neurology Intensive Care Unit of Ankara City Hospital, taking into account the circadian cycle.The type of the research is the experimental model with pre-test and post-test control group.Ankara City Hospital has included the research population in the last year.

It will consist of 1593 patients between the ages of 65-85 who are hospitalized in the Neurology Intensive Care Unit.Experimental and control groups will be created with simple randomization in randomization.The data were obtained from the socio-demographic characteristics form and the sleep pattern form developed by the researcher.

will be collected with

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of the therapeutic touch applied to the sleep patterns of individuals aged 65-85 years with chronic diseases who are treated in the Neurology Intensive Care Unit of Ankara City Hospital, taking into account the circadian cycle.Research Hospitalization in Ankara City Hospital Neurology Intensive Care It will be done with individuals who have chronic diseases in the 65-85 age range. Research It is planned to be held between November 2021 and December 2022.Therapeutic touch will be applied to the patients selected in the experimental and control groups among the patients who meet the research criteria in the intensive care units. After this application, the sleep pattern changes in the patients will be evaluated.Therapeutic touch will be applied to the patients selected in the experimental and control groups among the patients who meet the research criteria in the intensive care units. After this application, sleep pattern changes in patients will be evaluated. In the analysis of the research, dependent groups t test andindependent groups t test, Mann Whitney U and Kruskal Wallis tests will be used in non-parametric cases

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 1.65-85 years
* Having a Chronic Disease
* The patient's hospitalization in the Neurology Intensive Care Unit

Exclusion Criteria:

* Not in the age range of 65-85 years
* Not being able to communicate (being intubated, having hearing impairment, etc.)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The effect of therapeutic touch applied to the experimental group on sleep | at the end of 1 week
  The experimental group will be given therapeutic touch applications before. The sleep patterns of the patients who are applied therapeutic touch for 1 week will be followed. Sleep patterns will be followed by researchers and nurses by recording sleep hours and filling out sleep pattern questionnaire questions.

SECONDARY OUTCOMES:
Determining the sleep pattern of the Control Group | At the and of 1 week
  No intervention will be made on the control group. Sleep patterns of the patients will be monitored for 1 week. Sleep patterns will be followed by researchers and nurses by recording sleep hours and filling out sleep pattern questionnaire questions.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Bayır, Principal Investigator — KTO Karatay University
Locations (1):
- Berna Bayır, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No